CLINICAL TRIAL: NCT04611828
Title: Optimizing Peripheral Sensory Stimulation to Induce Sleep Slow Waves
Brief Title: Slow-wave Enhancement in Adults Aged 30-49
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-0337 Sub-Study 2; A538900 (Other: UW Madison); SMPH\PSYCHIATRY\PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Sleep
Keywords: sleep; cognitive performance

STUDY DESIGN:
Masking Description: Participants will be blind to the device condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Philips SmartSleep Device (Experimental): Participants will be instructed to sleep wearing the SmartSleep device at home for eight weeks, which will include three (3) two-week periods, one each of the following (in randomized order):
  * continuous fixed interval (ITI): SmartSleep will provide 1 Hz, inter-tone interval stimulation continuous during deep sleep opportunities
  * block: SmartSleep will provide 5s ON versus 5s OFF,1Hz inter-tone interval stimulation
  * in-phase adjustable: SmartSleep will provide constant stimulation with tones timed to be delivered during each upstate of the slow wave
  Between periods 1 and 2 and between periods 2 and 3, subjects will undergo one week of sham condition during which SmartSleep will record EEG during sleep using a no-volume sham stimulation
  Interventions: Device: Philips SmartSleep

INTERVENTIONS:
Device: Philips SmartSleep — closed-loop auditory stimulation

SUMMARY:
A single-site, randomized study to assess the effectiveness of different types of closed-loop auditory stimulation on slow-wave enhancement using SmartSleep in an astronaut-like sample of adults between the ages of 30 and 55. Secondary analyses will be performed to determine whether slow-wave enhancement influences neurobehavioral performance in this population. Participants will be on study for 8 weeks.

DETAILED DESCRIPTION:
The investigators seek to determine the extent to which various closed-loop auditory stimulation protocols (continuous fixed interval, block, in-phase adjustable) differentially affect slow-wave sleep. Participants will run the study for eight weeks, which includes wearing the SmartSleep device nightly, and completing one 3-min and one 20-min cognitive assessment battery each day, as well as computerized post-sleep questionnaires each morning, sleepiness scales three times a day, and a weekly evaluation of device comfort. This study will employ various types of auditory stimulation in order to determine 1) which stimulation pattern is maximally effective at enhancing slow wave activity (SWA) and 2) to assess cognitive performance associated with each stimulation algorithm. The study requires a longer duration so that sufficient data on each distinct type of stimulation may be collected.

Participants will be instructed to wear the SmartSleep device at home for three two-week periods, and will complete 10 nights per period of continuous fixed interval, block, or in-phase adjustable stimulation (in randomized order). Between each of these periods, participants will complete one week of sham condition (this condition records sleep EEG without any stimulation and is used to define each participant's typical sleep). During all eight weeks, participants will complete a 20-minute cognitive assessment in the evening, a five-minute cognitive assessment in the morning, and respond to the Karolinska Sleepiness Scale three times per day. The cognitive assessments will be accompanied by short questionnaires. Participants will receive text message reminders from study staff when it is time to perform these assessments.

Primary objective: Determine which stimulation type (e.g., Block stimulation, Fixed ITI, in-phase) is most effective at enhancing slow-waves slow-wave sleep relative to baseline sleep in a group of astronaut-like subjects in an ecologically valid setting.

Main secondary objective: Determine the extent to which various closed-loop auditory stimulation protocols (continuous fixed interval, block, inphase adjustable) differentially affect various aspects of neurobehavioral function using a set validated cognitive tasks as part of the Cognition battery.

Other secondary objectives: Explore the relationships between improvements in SWA and measures of subjective sleepiness as assessed by the Karolinska Sleepiness Scale

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Able to understand and speak English
* Left or right-handed participants may be included
* Participants have access to a cell phone that can receive text message reminders from study staff
* Participants have self-reported sleep latency (time taken to fall asleep) > 30 minutes no more than once per week
* Participants have self-reported wake time after sleep onset ≤ 30 minutes
* Participants with Body Mass Index (BMI) < 35 kg/m2 AND
* Participants self-report using an alarm to wake up ≥ 5 days a week
* Participants self-report sleeping one or more hours longer on weekends (or when given the opportunity) than they do on a typical work night

Exclusion Criteria:

* Participants who self-report taking medications that could affect sleep patterns
* Participants who have had travel in the last 2 weeks or who intend to travel during the experimental weeks with time zone shifts >3h
* Participants unlikely to comply with the protocol (e.g., uncooperative attitude)
* Individuals who self-report a current severe or chronic medical condition or sleep disorder that may affect sleep patterns
* Individuals who self-report a history of recurrent seizures or epilepsy or family history of hereditary epilepsy or have a history of medical conditions that could increase the chance of seizures (e.g. stroke, aneurysm, brain surgery, structural brain lesion)
* Participants who report not being consistent in their daily use of alcohol, caffeine, or nicotine
* Participants who are pregnant
* Participants who are night shift workers
* Individuals who self-report severe contact dermatitis or allergy to silicone, nickel or silver
* Individuals who self-report moderate hearing loss
* Self-reported history of excessive alcohol intake- selfreport > 21 drinks / wk or binge alcohol consumption ( >5 drinks per day)
* Excessive caffeine consumption (> 7 cups) combining all caffeinated drinks regularly absorbed during workdays. Caffeine intake must be regular and maintained throughout study and on testing days
* Participants who do not have internet access at home
* Participants who express unwillingness to forego napping on weekdays during the study
* Participants who smoke
* Participants with high risk of Obstructive Sleep Apnea (OSA) based on STOP-BANG Questionnaire ("yes" on at least 4 of 8 questions)
* High Risk of Restless Legs Syndrome (RLS) based on the short form Cambridge-Hopkins Screening questionnaire
* High Risk of Insomnia based on Insomnia Severity Index (score of 22 or higher)

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Slow Wave Activity between Audio Stimulation Condition and Sham Condition | up to 8 weeks
  To compare the three different types of stimulation, a common outcome was selected which is the change in slowwave activity between periods where the stimulation is applied versus equivalent periods, in a sham condition, where the stimulation is not applied but would have been applied. Three different conditions defined in the arm description will be measured: continuous fixed interval, block, and in-phase adjustable; each compared to the sham condition. Participant is blinded to each condition; all data collected over 8 weeks.

SECONDARY OUTCOMES:
Global Cognition Battery Score per Stimulation Condition | up to 8 weeks
  Cognition is a brief electronic battery that assesses several domains of cognitive function including attention, executive function, reaction time, short-term memory, working memory, spatial ability, and risk taking. Performance will be assessed under each stimulation condition and sham to determine whether enhancement impacts global performance. Total range of possible scores 10-100 where higher scores indicate increased cognition.
Karolinska Sleepiness Scale Score | up to 8 weeks
  These scales will be analyzed for changes in subjective sleepiness and perceived sleep quality between periods of different types of auditory stimulation and sham condition. Participants will be assessed 3 times daily (morning, afternoon, and evening), they will rate their alertness on a scale of 1 (extremely alert) to 9 (extremely sleepy, fighting sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Tononi, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT04611828/ICF_000.pdf